CLINICAL TRIAL: NCT01767883
Title: Improving Evidence-Based Primary Care for Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Family Physicians (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University at Buffalo (Other); University of Colorado, Denver (Other); National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAFP-CKD-102020846; 1R01DK090407-01A1 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Chronic Kidney Disease; Chronic Kidney Insufficiency; Chronic Renal Diseases; Chronic Renal Insufficiency; Kidney Insufficiency, Chronic
Keywords: Chronic Kidney Disease; CKD; TRANSLATE; Practice Facilitation; Practice-based research; CKD Guidelines
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Compact Disks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Facilitated Clinical Decision Support (Experimental): The primary care practices in this arm will receive:
  * CKD decision support algorithms added to their Clinical Decision Support
  * System Academic detailing concerning the rationale for the algorithms
  * On-going mentoring and practice facilitation
  Interventions: Other: Facilitated Clinical Decision Support
- Clinical Decision Support Only (Active Comparator): The primary care practices in this arm will receive:
  * CKD decision support algorithms added to their Clinical Decision Support System
  * Academic detailing concerning the rationale for the algorithms
  Interventions: Other: Clinical Decision Support Only

INTERVENTIONS:
Other: Facilitated Clinical Decision Support — The primary care practices in this arm will receive:
  * CKD decision support algorithms added to their Clinical Decision Support
  * System Academic detailing concerning the rationale for the algorithms
  * On-going mentoring and practice facilitation
  * Audit and feedback during quarterly reviews of practice data with the practice facilitator by videoconference.
  Other Names: Facilitated CDS,; CDS plus facilitation
  Arms: Facilitated Clinical Decision Support
Other: Clinical Decision Support Only — * CKD decision support algorithms added to their Clinical Decision Support
  * System Academic detailing concerning the rationale for the algorithms
  Other Names: CDS Only; "Comparator"
  Arms: Clinical Decision Support Only

SUMMARY:
Background: Chronic Kidney Disease (CKD) is under-recognized and under-treated in primary care offices and primary care physicians are generally not familiar with treatment guidelines. Even when diagnosed properly, as a chronic condition CKD is frequently associated with co-morbidities that make effective treatment difficult due to complexity of care. Availability of Clinical Decision Support (CDS) for CKD may help promote effective, evidence-based care, but evidence suggests that CDS alone may not be sufficient for quality improvement and other interventions such as CDS plus practice facilitation may be needed.

Purpose: The project aims to: 1) assess the viability of CDS in implementing evidence-based guidelines for Primary Care Practices (PCPs) and 2) to develop evidence-based practice guidelines that PCPs may use to enhance the care they provide to a difficult to manage segment of the healthcare population.

Methods: This is a randomized controlled trial of point-of-care CDS plus full TRANSLATE model of practice change, versus CDS alone. The study aims to analyze differences in promoting evidence-based care in primary care practices. Thirty-six practices will be recruited for this study. Patient inclusion criteria: adult patients with estimated Glomerular Filtration Rate (eGFR) of <60 and >15ml/min/1.73m2 confirmed with repeat testing over three or more months. A process evaluation will be conducted between the CDS practices with facilitation and the CDS only practices to assess clinical outcomes of CKD progression and all-cause mortality. Lastly, a cost-effective analysis will compare the cost-to-benefit ratio of CDS alone to that of CDS plus TRANSLATE (i.e. practice facilitation) in relation to cost per quality adjusted years of life. This study is funded by NIH NIDDK under R01 mechanism starting on 07/01/2011 and ending on 06/30/2016.

DETAILED DESCRIPTION:
The proposed trial tests the extent to which CDS plus facilitation promotes evidence-based care and improves the clinical outcomes of reduced disease progression and mortality in primary care practices. We also conduct an observational comparative effectiveness analysis of data from a larger database of electronic medical records in order to identify the most successful components of evidence-based care with respect to disease progression and all-cause mortality.

Specific Aim 1: Conduct a group randomized controlled trial of point-of-care computer decision support plus the full TRANSLATE model of practice change, versus computer decision support alone in promoting evidence-based care in primary care practices for all patients with an eGFR <60 and > 15 ml/min/1.73m2 confirmed with repeat testing over three or more months. (CKD stages 3 and 4) Hypothesis 1.1: CDS practices using the TRANSLATE model will provide a greater degree of evidence-based guideline-concordant care for CKD than CDS only practices.

Specific Aim 2: Conduct an intent-to-treat and process analysis between the CDS practices with facilitation versus the CDS only practices of the clinical outcomes of CKD progression and all-cause mortality.

Hypothesis 2.1: Patients with stage 3 and 4 CKD in facilitated practices will have slower CKD progression than patients in CDS only practices.

Hypothesis 2.2: Patients with stage 3 and 4 CKD in facilitated practices will have significantly lower all-cause mortality than stage 3 and 4 patients in CDS only practices.

Hypothesis 2.3: The process evaluation will determine through qualitative methods the fidelity of the facilitated TRANSLATE program; find the challenges and enablers of the implementation process, the role of facilitation, and the contextual factors that contribute to TRANSLATE decisions and strategies; and translate lessons learned into pragmatic "best practices" for future facilitation and dissemination.

Specific Aim 3: Conduct a cost-effectiveness analysis that will compare the benefit of the intervention of computer decision support alone against the intervention of computer decision support plus TRANSLATE (practice facilitation). Hypothesis 3.1 The intervention of computer decision support plus TRANSLATE is more cost-effectiveness than the intervention of computer decision support alone.

ELIGIBILITY:
Inclusion Criteria:

* all individuals whose primary care provider offices participate in the study who is over the age of 18 with a diagnosis of stages 2-4 of CKD and/or diabetes and/or hypertension and/or one eGFR <60 and/or one urine albumin/creatinine ratio >30

Exclusion Criteria:

* individual patients whose primary care provider's practice has not signed practice and data use agreements with the AAFP NRN to participate in this practice improvement project at the practice level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27000 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Degree of evidence-based guideline-concordant care for CKD | up to 3 years
  Percentage of patients at goal for:
  Control Blood Pressure Control LDL Control HbA1C Use ACE/ARB Eliminate NSAID/Cox-2 use Refer to Nephrologist Eliminate Smoking

SECONDARY OUTCOMES:
CKD Management Process Measures | upt to 3 years
  Percentage of patients who have:
  Diagnosis of CKD Annual Microalbumin/Creatinine Ratio Annual LDL Annual A1c Follow up creatinine measure Follow up ACR measure
Cost of intervention | up to 3 years
  Extra costs of the "Translate CKD" intervention and the control intervention, compared to no intervention. Claims data from Centers for Medicare & Medicaid Services, additional practice and patient costs
All-cause mortality | up to 3 years
  Death data from the CDC National Death Index

OTHER OUTCOMES:
Process evaluation outcomes | Change from Baseline practice performance at 3 years
  Qualitative and descriptive measure of practice performance, physician and staff satisfaction and process changes as obtained through site visit observations, interviews and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Chester H Fox, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- American Academy of Family Physicians, Leawood, Kansas, United States

REFERENCES:
- [Derived] Carroll JK, Pulver G, Dickinson LM, Pace WD, Vassalotti JA, Kimminau KS, Manning BK, Staton EW, Fox CH. Effect of 2 Clinical Decision Support Strategies on Chronic Kidney Disease Outcomes in Primary Care: A Cluster Randomized Trial. JAMA Netw Open. 2018 Oct 5;1(6):e183377. doi: 10.1001/jamanetworkopen.2018.3377. PMID 30646261
- [Derived] Loskutova NY, Smail C, Ajayi K, Pace WD, Fox CH. Recruiting primary care practices for practice-based research: a case study of a group-randomized study (TRANSLATE CKD) recruitment process. Fam Pract. 2018 Jan 16;35(1):111-116. doi: 10.1093/fampra/cmx064. PMID 28985294
- [Derived] Cipparone CW, Withiam-Leitch M, Kimminau KS, Fox CH, Singh R, Kahn L. Inaccuracy of ICD-9 Codes for Chronic Kidney Disease: A Study from Two Practice-based Research Networks (PBRNs). J Am Board Fam Med. 2015 Sep-Oct;28(5):678-82. doi: 10.3122/jabfm.2015.05.140136. PMID 26355142
- [Derived] Kahn LS, Vest BM, Madurai N, Singh R, York TR, Cipparone CW, Reilly S, Malik KS, Fox CH. Chronic kidney disease (CKD) treatment burden among low-income primary care patients. Chronic Illn. 2015 Sep;11(3):171-83. doi: 10.1177/1742395314559751. Epub 2014 Nov 21. PMID 25416418
- [Derived] Fox CH, Vest BM, Kahn LS, Dickinson LM, Fang H, Pace W, Kimminau K, Vassalotti J, Loskutova N, Peterson K. Improving evidence-based primary care for chronic kidney disease: study protocol for a cluster randomized control trial for translating evidence into practice (TRANSLATE CKD). Implement Sci. 2013 Aug 8;8:88. doi: 10.1186/1748-5908-8-88. PMID 23927603